CLINICAL TRIAL: NCT06760871
Title: The Effect of Cold Steam Application on Nausea and Vomiting After Laparoscopic Abdominal Surgery: Randomized Controlled Trial
Brief Title: The Effect of Cold Steam Application on Nausea and Vomiting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeynep Kızılcık Ozkan, associate professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 358/2024
Record Dates: First submitted 2024-12-17; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group will receive inhaled cold vapour. Patients in the control group will not be intervened within the scope of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will receive inhaled cold vapour.
  Interventions: Other: nebulised distilled water
- Control group (No Intervention): Patients in the control group will not be intervened within the scope of the study.

INTERVENTIONS:
Other: nebulised distilled water — After the surgery, the patients will be admitted to the ward and taken to the bed, and their care and treatment will be applied by the nurse. Afterwards, the researcher will apply cold vapour as an inhaler for 15 minutes. For this application, the stand to which the ultrasonic nebuliser device is connected will be positioned close to the patient's bed. 200 ml of distilled water will be placed in the liquid reservoir of the device. The patient will be given a comfortable position and the device will be adjusted so that the steam hose covers the patient's mouth and nose and the patient will be allowed to inhale the steam through the mouth and nose. After the electrical connection of the device is provided, the device will be started and cold steam application will begin. In the 1st hour, inhaler cold water vapour application will be performed for 15 minutes.
  Arms: Experimental group

SUMMARY:
The aim of this study was to determine the effect of cold vapour applied to patients undergoing laparoscopic abdominal surgery primarily on nausea and vomiting and secondarily on antiemetic requirement, patient satisfaction and thirst.

H1: Cold steam application after surgical intervention has a decreasing effect on postoperative nausea.

H2: Cold steam application after surgical intervention has a decreasing effect on postoperative vomiting.

H3: Cold steam application after surgical intervention reduces the need for antiemetic drugs.

H4: Cold steam application after surgical intervention has a satisfactory effect on reducing nausea and vomiting.

DETAILED DESCRIPTION:
The research will be conducted with the participation of surgical patients who underwent laporoscopic abdominal surgery between December 2024 and March 2025 in the General Surgery Department of Trakya University Hospital.

Effect size of 0.2 was predicted, the smallest possible significant correlation coefficient between repeated measurements was accepted as 0.3, and the minimum number of people to be included in the sample was calculated as 80, consisting of 40 patients from each group with a 95% confidence level, 5% margin of error and 80% power value. In case of possible data loss, drop out rate was accepted as 10% and 44 patients were included in each group.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing abdominal surgery under general anaesthesia,
* Admitted to the general surgery ward after surgery,
* Who volunteered to participate in the research,
* No mental disability,
* 18 years of age,
* Literate,
* Accepting random selection,
* without Turkish communication problems,
* No preoperative oncological treatment,
* undergoing elective surgery,
* Postoperatively without a nasogastric catheter,
* with an operation time <4 hours,
* Laparoscopic surgery performed,
* No postoperative nausea and vomiting or mild/moderate nausea,
* Patients with ASA score 1, 2 or 3 were determined as inclusion criteria.

Exclusion Criteria:

* Severe nausea or active vomiting prior to administration,
* Migraine, vertigo, etc. who may experience nausea and vomiting due to vestibular disease, pregnancy,
* COPD, asthma, etc. with respiratory problems,
* Not accepting the application of cold steam,
* Not accepting random selection,
* Those with a history of chemotherapy or radiotherapy before surgery,
* Patients who underwent sudden movement changes (bed change, patient transfer, etc.) during the data collection period (0 to 2nd hour),

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
nausea rate | 6 months
  Nausea rate (%)

SECONDARY OUTCOMES:
Antiemetic requirement | 6 months
  Antiemetic requirement (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Hospital, Edirne, Turkey (Türkiye)